CLINICAL TRIAL: NCT02945878
Title: Predictive Factors of Acute Oral Mucositis Induced by Intensity-Modulated Radiation Therapy With Concurrent Chemotherapy for Local Advanced Nasopharyngeal Carcinoma
Brief Title: Predictive Factors of Acute Oral Mucositis Induced by Chemo-radiotherapy for Local Advanced Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NPC-MUCO
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2016-10

CONDITIONS: Nasopharyngeal Neoplasms; Stomatitis
Keywords: radiotherapy, oral mucositis,oral mucosa protection
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Stomatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective, observational study to analyze the clinical and dosimetric factors about the radiation oral mucositis caused by radical chemo-radiotherapy for nasopharyngeal carcinoma patients and try to find the indicators for acute radiation oral mucositis.

DETAILED DESCRIPTION:
All patients received 1 - 3 concurrent chemotherapy during the intensity modulated radiotherapy. Before radiotherapy, three types of mouth mucosa are contoured in all treatment plans. Oral mucosa grades are recorded before and during treatment. Dose-volume Histograms are got to analyze the associated factors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically conformed Initial nasopharyngeal carcinoma
2. Patients can feed through the mouth.
3. ECOG (Eastern Cooperative Oncology Group) : 0-1.
4. No history of chemo-radiotherapy, immuno-therapy or biotherapy.
5. Normal hemodynamic indices before the recruitment (including white blood cell count>4.0×109/L, neutrophil count>1.5×109/L, platelet count >100×109/L, hemoglobin≥90g/l, normal liver/kidney function).
6. Informed consent signed.

Exclusion Criteria:

1. History of malignant tumors.
2. Any severe complications contraindicated chemotherapy or radiotherapy.
3. Medical history of central nervous system, cognitive or psychological diseases;
4. Pregnant or nursing women.
5. Patients with mental disease cannot complete the questionaire.
6. Patients refused the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically conformed Initial nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
gradings of oral mucositis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Chen, Professor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No